CLINICAL TRIAL: NCT04910594
Title: Prospective, Open-label, Multicenter Clinical Study for the Efficacy and Safety of Recombinant Human Erythropoietin in the Treatment of Anemia in Patients With Lymphoma
Brief Title: Clinical Study the Efficacy and Safety of Rh-EPO in the Treatment of Anemia in Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First People's Hospital of Hangzhou (Other); Zhejiang Provincial Tongde Hospital (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Zhejiang Cancer Hospital (Other); Wenzhou Central Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Affiliated Hospital of Jiaxing University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0135
Record Dates: First submitted 2021-05-31; First posted 2021-06-02 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-05

CONDITIONS: Lymphoma; Anemia
Keywords: lymphoma; anemia; recombinant human erythropoietin
MeSH Terms: conditions — Lymphoma; Anemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: recombinant human erythropoietin — To determine the efficacy and safety of recombinant human erythropoietin in improving anemia in patients with lymphoma, and to improve the quality of life and the efficacy of chemotherapy in patients with lymphoma.
  Other Names: EPO

SUMMARY:
The incidence of lymphoma and anemia is high and the clinical harm is great.However, it has not yet attracted enough clinical attention, and domestic rHuEPO (trade name: Ebio).Shenyang Sansheng Pharmaceutical Co., Ltd.) for lymphoma and anemia patients are less clinical studies.Therefore, a prospective, open-label, multicenter clinical study of recombinant human erythropoietin in the treatment of anemia in patients with lymphoma is planned to analyze the efficacy and safety of recombinant human erythropoietin in patients with lymphoma and anemia, so as to determine the clinical benefits of recombinant human erythropoietin in patients with lymphoma and anemia.

DETAILED DESCRIPTION:
Anemia is a common complication of malignant lymphoma.Approximately 30-40% of lymphoma patients develop anemia before chemotherapy begins [1].Common clinical manifestations of anemia include fatigue, weakness, dizziness, headache, shortness of breath, depression and other symptoms.Lymphoma anemia has a complex etiology, including chronic anemia (ACD), autoimmune hemolytic anemia (AIHA), bone marrow infiltration, malnutrition, and blood loss [2].

The incidence and prevalence of anemia are positively correlated with the severity of the disease and the chemotherapy cycle.A multi-center survey of anemia in patients with lymphoma in Shanghai published in 2020 included 501 patients, and the results showed that the incidence of anemia in patients with lymphoma was 35.5%;The prevalence of anemia was 62.7 percent during the entire 6-month follow-up period.Among the newly treated patients, the incidence of anemia was significantly higher in patients with Ann Arbor staging from Ⅲ to normal (P < 0.001), indicating that the incidence of anemia was related to the severity of the disease.In addition, chemotherapy is also a key factor in the development of anemia during the course of the disease.In this Shanghai survey, 267 newly treated lymphoma patients receiving chemotherapy increased the rate of newly diagnosed anaemia from 6.82% in the first course of chemotherapy to 43.18% in the fourth course of chemotherapy and above [3].The results of the European Anemia Survey of 15,367 cancer patients (ECAS) conducted in 2004 also showed a high incidence of anemia in lymphoma patients (2 260 lymphoma patients, 52.5%) [4], and the cumulative incidence of anemia in patients increased with the increase of chemotherapy cycles [5].

Anemia can reduce the quality of life of tumor patients, affect the therapeutic effect, and shorten the survival period of patients [6].A number of studies have shown that anemia is an independent risk factor affecting the prognosis of patients with diffuse large B-cell lymphoma (DLBCL) [7, 8].Compared with patients with Hb≥10 g/dL, those with Hb≥10 g/dL were more likely to have bone marrow involvement before treatment.Patients with lymphoma at 10 g/dL showed a lower event-free and disease-free survival.R-CHOP regimen (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone) was also an independent predictor of disease recurrence and an independent predictor of International Prognostic Index (IPI) 6 months after chemotherapy [7].After 3-4 courses of chemotherapy, the efficacy of newly treated lymphoma patients was evaluated, and it was found that the efficacy gradually deteriorated with the increase of anemia level [3].Another domestic study found that among 12L patients treated with R-CHOP regimen, 77 patients had grade 2 anemia or above (Hb < 10g/ dL, 63.6%), and the analysis results of the relationship between different Hb grades and overall survival showed that the greater the degree of anemia, the lower the overall survival rate of patients [9].

Although patients with lymphoma have a higher incidence of anemia, most patients do not receive prompt treatment.ECAS survey showed that anemia treatment rate of lymphoma patients was low, only 47.4%[4].For patients with tumor-associated anemia, treatment includes red blood cell transfusions, erythropoiesis stimulants (ESAs), and iron.Before the emergence of ESAs, blood transfusion was the main treatment.Although blood transfusions can quickly raise Hb levels, there are risks associated with allergies, viral infection, immunosuppression and iron overload.So the only Hb<Blood transfusion should be considered at 60 g/L or when hypoxia is urgently corrected clinically.ECAS survey showed that recombinant human erythropoietin (rHuEPO) was the main treatment for cancer anemia, but the treatment rate was low (17.4%) [4].Previous studies have confirmed that rHuEPO has achieved positive efficacy in the treatment of anemia caused by solid tumors and hematologic tumors.A 2008 study showed that the response rate of 33 NHL patients receiving chemotherapy treated with rHuEPO was 84.8%, and the earlier the treatment of rHuEPO, the higher the response rate [10].Glossmann J P et al. investigated the effects of rHuEPO on Hb level, blood transfusion volume and quality of life in patients with recurrent lymphoma, and found that while rHuEPO increased Hb level, it reduced the need for blood transfusion and improved the quality of life of patients [11].However, in recent years, concerns about the safety of rHuEPO in cancer patients have limited its clinical application.In recent years, large meta-analyses and randomized controlled studies have not shown that ESAs promote tumor progression [12-15].The "Management of Anemia and Iron Deficiency in Cancer Patients: ESMO Clinical Practice Guidelines" published by the European Society of Physicians of Oncology (ESMO) in 2018 also clearly pointed out that the standardized use of ESAS would not promote the progression or recurrence of cancer disease [16].Therefore, the appropriate use of rHuEPO in lymphoma patients undergoing chemotherapy can provide clinical benefits such as reduced need for blood transfusion and improved quality of life without excessive safety concerns.

In view of the high incidence of lymphoma anemia and greater clinical harm.However, it has not yet attracted enough clinical attention, and domestic rHuEPO (trade name: Ebio).Shenyang Sansheng Pharmaceutical Co., Ltd.) for lymphoma and anemia patients are less clinical studies.Therefore, a prospective, open-label, multicenter clinical study of recombinant human erythropoietin in the treatment of anemia in patients with lymphoma is planned to analyze the efficacy and safety of recombinant human erythropoietin in patients with lymphoma and anemia, so as to determine the clinical benefits of recombinant human erythropoietin in patients with lymphoma and anemia.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological diagnosis: lymphoma;
2. Age 14 to 65, no gender limitation;
3. ECOG physical condition score was 0~3;
4. Life expectancy >6 months;
5. did not receive recombinant human erythropoietin treatment within 30 days before the first day;
6. Complete liver and kidney function (creatinine ≦1.5*ULN, BUN≦1.5*ULN, ALT≦2*ULN, AST≦2*ULN, total bilirubin ≦1.5*ULN;ULN: upper limit of normal value);
7. Willing to sign the informed consent, can understand and abide by the requirements of the study.

Exclusion Criteria:

1. Active infections requiring intravenous antibiotic treatment and any active malignancies (except lymphomas);
2. Grade III or IV heart failure, uncontrolled hypertension or hypotension, and associated risk or event of thromboembolism;
3. Severe hepatic and renal insufficiency;
4. Patients who have received radiotherapy or chemotherapy for other tumors (except lymphoma) within 6 months;
5. other anemia diseases (such as aplastic anemia, thalassemia, myelodysplastic syndrome, etc.);
6. Inability to understand and follow the study protocol or inability to sign the informed consent.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-02-14 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin response rate of subjects during treatment. | up to 20weeks
  A hemoglobin response was defined as an increase in hemoglobin levels of ≥ 1.0 g/dL from baseline during 2 or more consecutive assessments (2 weeks apart) without red blood cell infusion.

SECONDARY OUTCOMES:
The time of the first hemoglobin response | up to 20weeks
  The time of the first hemoglobin response

CONTACTS AND LOCATIONS:
Overall Officials: wenbin qian, Principal Investigator — 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hanzhou, China

IPD SHARING:
Plan to Share IPD: Yes
share the dates when published
Supporting Information: Study Protocol, CSR
Time Frame: up to ten years
Access Criteria: by pubmed